CLINICAL TRIAL: NCT02967991
Title: 19 Versus 22-Gauge Fine Needle Biopsy (FNB) Needles for Endoscopic Ultrasound Guided Liver Biopsy (EUS-LB): A Prospective Pilot Study
Brief Title: 19 Versus 22-Gauge Needle for EUS-LB
Acronym: EUSLB1922
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016-0281
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-06

CONDITIONS: Diagnoses Diseases; Ultrasound Therapy; Complications; Liver Diseases
Keywords: EUS; Biopsy; Liver; FNA; FNB
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 19 Left (Active Comparator): EUS-guided liver biopsy using a19-gauge liver biopsy in the left lobe
  Interventions: Device: EUS-guided liver biopsy
- 22 Left (Experimental): EUS-guided liver biopsy using a 22-gauge liver biopsy in the left lobe
  Interventions: Device: EUS-guided liver biopsy
- 19 Right (Active Comparator): EUS-guided liver biopsy using a 19-gauge liver biopsy in the right lobe
  Interventions: Device: EUS-guided liver biopsy
- 22 Right (Experimental): EUS-guided liver biopsy using a 22-gauge liver biopsy in the right lobe
  Interventions: Device: EUS-guided liver biopsy

INTERVENTIONS:
Device: EUS-guided liver biopsy — Endoscopic ultrasound guided liver biopsy

SUMMARY:
Chronic liver disorders (CLD) are a major cause of morbidity and mortality for individuals in the US. Though serologic analysis will often lead to a conclusive diagnosis, liver biopsy remains an important method for helping to determine the etiology and stage of LD. Percutaneous liver biopsy (PLB), transjugular liver biopsy (TLB) and surgical liver biopsy (SLB) are alternative methods for obtaining hepatic tissue. In recent years endoscopic ultrasound guided-liver biopsy (EUS-LB) has come to the forefront as a safe and effective method for obtaining tissue in CLD. There are several studies of the safety of EUS-LB as well as the adequacy of specimens obtained in this fashion. Most studies involve a 19-gauge needle, therefore in this study the investigators hope to compare the tissue yields of a 22-gauge fine needle biopsy (FNB) needle, in comparison to conventional 19-gauge. The investigators predict that 19 and 22 gauge FNB needle will demonstrate similar diagnostic accuracy, with less visible blood artifact. Similarly the investigators predict the safety to be equal.

DETAILED DESCRIPTION:
3 BACKGROUND AND SIGNIFICANCE Chronic liver disease has a number of causes, and leads to significant mortality and morbidity in the United States. It has been estimated that roughly 36,000 individuals die annually from the burden of chronic liver disease, thus early diagnosis and intervention are paramount to preventing such complications. Though serologic markers and non-invasive diagnostic imaging modalities are used as a method for determining the underlying disease process, these methods lack the specificity of determining etiology of a patient's chronic liver disease. Therefore, liver biopsy remains the "gold standard" for obtaining valuable diagnostic and prognostic information.

At present there exist several methods for liver tissue acquisition. The most widely accepted method remains percutaneous route (PLB), which utilizes percussion or imaging to localization the biopsy site. The issue with this approach is its potential complication of post-procedural pain in up to 84%, bleeding in 1/2500-10,000 procedures, with under 1/10,000 of these cases being fatal. Another means for obtaining tissue samples is the transjugular route (TLB), which also allows for portal pressure measurement, and is usually reserved for patients with coagulopathy.

More recently, endoscopic ultrasound guided liver biopsy (EUS-LB) has been developed as a newer LB technique. The feasibility of EUS-LB for liver lesions has been validated yielding excellent diagnostic results in several studies. This technique has also been evaluated for hepatic parenchymal disease with up to 90% diagnostic yield. Subsequently, EUS-LB using a 19-gauge needle was compared to percutaneous/transjugular routes showing at least comparative, and in some instances improved sample acquisition, versus other methods. Different 19-gauge needles have been utilized in this setting yielding variable diagnostic specimens. However, there has yet to be comparison of 19 versus a 22-gauge core biopsy needle for EUS-LB. The safety profile with the 19g needle is remarkably good; it seems logical that a smaller needle would be at least as good, if not better.

Primary End Points

1. Proportion of cases for which a histologic diagnosis could be made based upon the amount of tissue obtained with the needle (using total portal structures > 5 or length of the longest piece (LLP) > 15 mm).
2. Number of portal tracts (PT) in the specimen
3. Aggregate specimen length (ASL), length of the longest piece (LLP), and degree of fragmentation Secondary End Points

1. Presence of a visible core specimen 2. Presence of visible clots in specimen 3. Adverse events (AE) and serious adverse events (SAE) 4 HYPOTHESIS AND SPECIFIC aims

4.1 Hypothesis The investigators predict that the 19-gauge needle and 22-gauge core needle will have similar ability to obtain adequate EUS-LB specimens 4.2 Specific Aim 1 To determine the adequacy of EUS-LB using a 22-gauge core needle as compared with 19-gauge needle 4.3 Specific Aim 2 To determine if the 22-gauge core needle will demonstrate less blood artifact during the time of EUS-LB as compared with 19-gauge needle.

6 STUDY DESIGN 6.1 Description This is a prospective trial comparing the biopsy specimen adequacy of 19 versus 22-gauge core needle for EUS-LB.

6 6.3 Recruitment Patients shall be recruited in the pre-procedural endoscopy area. After identifying subjects, a study investigator shall discuss the study in detail either in person (at which point the patient will read the consent form). A second individual will witness the consent.

6.4 Study Duration 6.4.1 Approximate Duration of Subject Participation Participation in this study is until 1 week post-procedure. 6.4.2 Approximate Duration of Study The duration of the study shall last until 6 months from enrollment of the last study participant. This shall allow for analysis of final data points and construction of a manuscript.

6.5 Procedures Epic electronic health records database will allow for availability of demographic data and office-based follow-up records. Provation MD software information will provide details regarding endoscopic parameters and intervention performed.

Electronic records gathered for study purposes will only be available to study investigators and will be stored on an encrypted hard drive on a computer. Data will initially be entered with protected health information (PHI) attached so that all information can be obtained. Once all data collection is complete identifiers will be removed and random number assigned to the patients.

Paper copies of study questionnaires will be filled out in the endoscopy center and stored in a locked cabinet in the endoscopy center workroom. The door to the workroom with the cabinet is locked after hours and the endoscopy center is locked after hours as well.

Upon initial encounter, the study shall be described to the patient in detail by one of the study investigators and informed consent obtained.

Once the patients has agreed to participate, demographic data will be obtained including; age, gender, height [inches (in)], weight [pounds (lb)], body mass index (BMI)(lb/in2), past medical history [in particular diagnosis of liver disease, biliary or pancreatic disease, ascites, encephalopathy, portal hypertension, portal hypertension-related bleeding (ie. varices), liver cancer or masses]. Past surgical history shall be obtained regarding prior cholecystectomy, hepatobiliary or pancreatic surgery (i.e. pancreaticojejunostomy) or bariatric surgery (ie. Roux-en-Y gastric bypass). Medication and social history shall be performed regarding alcohol intake per week and hepatotoxic medications (i.e. acetaminophen). A baseline INR and platelet count shall be performed on all individuals prior to EUS-LB, as is the standard of care.

EUS-LB Protocol

Patients undergoing EUS-LB receive sedation prior to the procedure, as per normal practice. This is provided by a certified registered nurse anesthetist (CRNA). The endosonographic study will be conducted with a linear array echoendoscope (GF-UC140-AL5; Olympus America, Center Valley, PA). Before needle puncture of the desired lobe, color Doppler imaging will be used to ensure the lack of vascular structures in the trajectory of the needle. The EUS-LB will be performed in widely separated regions of the liver using a 19-gauge EUS-FNA (fine needle aspiration) needle (Expect Flexible 19g, Boston Scientific, Marlborough, MA) and a 22-gauge FNB needle (SharkCore, Beacon Endoscopic, Sunnyvale, CA, or Acquire 22g, Boston Scientific, Marlborough, MA). A computer-generated randomized schema shall determine initial needle gauge selection.

The left lobe is described as liver parenchyma identified a few centimeters below the gastroesophageal junction with the echoendoscope torqued clockwise. The right lobe is consider the large area of liver tissue can be seen through the duodenal bulb, near the gallbladder. The stylet is removed, heparin flushed through the needle lumen, and the suction device set and attached to the needle hub. The prepared needle is then inserted into the echoendoscope, A transgastric approach will be used to obtain samples from the left lobe of the liver; a transduodenal approach, with the linear echoendoscope positioned in the duodenal bulb, will be used to obtain samples from the large amount of liver parenchyma seen in that location. Once adequate liver parenchymal penetration will be achieved with the needle (∼2-6 cm), full suction will be applied with a 20-mL vacuum syringe. One pass consists of a total of 7 to 10 to-and-fro needle motions with the fanning technique applied under direct and continuous endosonographic visualization of the tip of the needle.

The needle will then be removed from the echoendoscope. The specimen will be pushed from the needle with the stylet directly into a microsieve, and blood washed from the specimen with a gentle saline rinse. The endosonographer looks for multiple pieces of light brown tissue approximately 5 to 15 mm in length. The tissue cores are then "floated" off the microsieve into formalin solution. Then, a second pass will be made from the same region of the liver using the alternate needle used from the first pass. Heparin is flushed through the needle lumen prior to the next pass. The biopsy process is then repeated on the opposite liver lobe. Two passes per liver lobe are made; one with the standard 19g EUS-FNA needle, and one with the 22g EUS core needle. All patients are closely observed in the recovery area for 1 hour after the procedure, as per our standard policy. Patients will be followed-up with by a phone call the next day and at 1 week after the procedure.

Sample Processing The surgical pathology department, per a specific protocol for clinical practice, will process the EUS-LB samples. Tissue samples are left in formalin for at least 1 hour before processing. The contents of the formalin jar will be poured into a petri dish, and visible cores of liver tissue picked out with small forceps by the surgical pathology technician. These pieces are arranged in a linear fashion on lens paper, then the specimen photographed alongside a ruler to estimates pre-processing tissue lengths. Samples from both lobes and the different needles will be submitted for evaluation separately. The tissue will be processed in standard fashion, and slide blanks made (5-μm tissue thickness). These blanks are stained with hematoxylin and eosin, trichrome, and reticulin, with other special stains done as needed. The slides is digitized using a whole slide scanner (ScanScope CS; Aperio Technologies, Inc, Vista, CA), and the digitized images used for quantitative analysis (eSlide Manager; Aperio Technologies, Inc). Quantification of sample length (mm) and portal triads is performed by 2 of the investigators, annotating the digital images with the software. Fellowship-trained GI pathologists then perform histologic interpretation for clinical use.

Post-Procedural Follow-up After undergoing the procedure, patients will receive a 1week follow-up phone call to monitor for adverse events (i.e. bleeding).

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing EUS-LB
2. Platelet count > 50,000
3. International normalized ratio (INR) < 1.5
4. Age > 18 years
5. Non-pregnant patients

Exclusion Criteria:

1. Age < 18 years
2. Pregnant Patients
3. Inability to obtain consent
4. Anticoagulants or anti-platelet agents use (excluding aspirin) within the last 7-10 days
5. Platelet count < 50,000
6. INR > 1.5
7. Presence of ascites
8. Known liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Diehl, M.D., Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Rockey DC, Bissell DM. Noninvasive measures of liver fibrosis. Hepatology. 2006 Feb;43(2 Suppl 1):S113-20. doi: 10.1002/hep.21046. PMID 16447288
- [Background] Rockey DC. Noninvasive assessment of liver fibrosis and portal hypertension with transient elastography. Gastroenterology. 2008 Jan;134(1):8-14. doi: 10.1053/j.gastro.2007.11.053. PMID 18166342
- [Background] Ziol M, Handra-Luca A, Kettaneh A, Christidis C, Mal F, Kazemi F, de Ledinghen V, Marcellin P, Dhumeaux D, Trinchet JC, Beaugrand M. Noninvasive assessment of liver fibrosis by measurement of stiffness in patients with chronic hepatitis C. Hepatology. 2005 Jan;41(1):48-54. doi: 10.1002/hep.20506. PMID 15690481
- [Background] Sherlock S, Dick R, Van Leeuwen DJ. Liver biopsy today. The Royal Free Hospital experience. J Hepatol. 1985;1(1):75-85. doi: 10.1016/s0168-8278(85)80070-2. PMID 3902951
- [Background] Eisenberg E, Konopniki M, Veitsman E, Kramskay R, Gaitini D, Baruch Y. Prevalence and characteristics of pain induced by percutaneous liver biopsy. Anesth Analg. 2003 May;96(5):1392-1396. doi: 10.1213/01.ANE.0000060453.74744.17. PMID 12707140
- [Background] Perrault J, McGill DB, Ott BJ, Taylor WF. Liver biopsy: complications in 1000 inpatients and outpatients. Gastroenterology. 1978 Jan;74(1):103-6. PMID 618417
- [Background] Firpi RJ, Soldevila-Pico C, Abdelmalek MF, Morelli G, Judah J, Nelson DR. Short recovery time after percutaneous liver biopsy: should we change our current practices? Clin Gastroenterol Hepatol. 2005 Sep;3(9):926-9. doi: 10.1016/s1542-3565(05)00294-6. PMID 16234032
- [Background] Stone MA, Mayberry JF. An audit of ultrasound guided liver biopsies: a need for evidence-based practice. Hepatogastroenterology. 1996 Mar-Apr;43(8):432-4. PMID 8714240
- [Background] McGill DB, Rakela J, Zinsmeister AR, Ott BJ. A 21-year experience with major hemorrhage after percutaneous liver biopsy. Gastroenterology. 1990 Nov;99(5):1396-400. doi: 10.1016/0016-5085(90)91167-5. PMID 2101588
- [Background] Janes CH, Lindor KD. Outcome of patients hospitalized for complications after outpatient liver biopsy. Ann Intern Med. 1993 Jan 15;118(2):96-8. doi: 10.7326/0003-4819-118-2-199301150-00003. PMID 8416324
- [Background] Piccinino F, Sagnelli E, Pasquale G, Giusti G. Complications following percutaneous liver biopsy. A multicentre retrospective study on 68,276 biopsies. J Hepatol. 1986;2(2):165-73. doi: 10.1016/s0168-8278(86)80075-7. PMID 3958472
- [Background] Huang JF, Hsieh MY, Dai CY, Hou NJ, Lee LP, Lin ZY, Chen SC, Wang LY, Hsieh MY, Chang WY, Yu ML, Chuang WL. The incidence and risks of liver biopsy in non-cirrhotic patients: An evaluation of 3806 biopsies. Gut. 2007 May;56(5):736-7. doi: 10.1136/gut.2006.115410. No abstract available. PMID 17440193
- [Background] Cadranel JF, Rufat P, Degos F. Practices of liver biopsy in France: results of a prospective nationwide survey. For the Group of Epidemiology of the French Association for the Study of the Liver (AFEF). Hepatology. 2000 Sep;32(3):477-81. doi: 10.1053/jhep.2000.16602. PMID 10960438
- [Background] Myers RP, Fong A, Shaheen AA. Utilization rates, complications and costs of percutaneous liver biopsy: a population-based study including 4275 biopsies. Liver Int. 2008 May;28(5):705-12. doi: 10.1111/j.1478-3231.2008.01691.x. PMID 18433397
- [Background] Bravo AA, Sheth SG, Chopra S. Liver biopsy. N Engl J Med. 2001 Feb 15;344(7):495-500. doi: 10.1056/NEJM200102153440706. No abstract available. PMID 11172192
- [Background] Lebrec D, Goldfarb G, Degott C, Rueff B, Benhamou JP. Transvenous liver biopsy: an experience based on 1000 hepatic tissue samplings with this procedure. Gastroenterology. 1982 Aug;83(2):338-40. PMID 7084612
- [Background] Bull HJ, Gilmore IT, Bradley RD, Marigold JH, Thompson RP. Experience with transjugular liver biopsy. Gut. 1983 Nov;24(11):1057-60. doi: 10.1136/gut.24.11.1057. PMID 6629116
- [Background] Orlando R, Lirussi F, Okolicsanyi L. Laparoscopy and liver biopsy: further evidence that the two procedures improve the diagnosis of liver cirrhosis. A retrospective study of 1,003 consecutive examinations. J Clin Gastroenterol. 1990 Feb;12(1):47-52. PMID 2137481
- [Background] Poniachik J, Bernstein DE, Reddy KR, Jeffers LJ, Coelho-Little ME, Civantos F, Schiff ER. The role of laparoscopy in the diagnosis of cirrhosis. Gastrointest Endosc. 1996 Jun;43(6):568-71. doi: 10.1016/s0016-5107(96)70192-x. PMID 8781934
- [Background] Denzer U, Arnoldy A, Kanzler S, Galle PR, Dienes HP, Lohse AW. Prospective randomized comparison of minilaparoscopy and percutaneous liver biopsy: diagnosis of cirrhosis and complications. J Clin Gastroenterol. 2007 Jan;41(1):103-10. doi: 10.1097/01.mcg.0000225612.86846.82. PMID 17198072
- [Background] Stavropoulos SN, Im GY, Jlayer Z, Harris MD, Pitea TC, Turi GK, Malet PF, Friedel DM, Grendell JH. High yield of same-session EUS-guided liver biopsy by 19-gauge FNA needle in patients undergoing EUS to exclude biliary obstruction. Gastrointest Endosc. 2012 Feb;75(2):310-8. doi: 10.1016/j.gie.2011.09.043. PMID 22248599
- [Background] Diehl DL, Johal AS, Khara HS, Stavropoulos SN, Al-Haddad M, Ramesh J, Varadarajulu S, Aslanian H, Gordon SR, Shieh FK, Pineda-Bonilla JJ, Dunkelberger T, Gondim DD, Chen EZ. Endoscopic ultrasound-guided liver biopsy: a multicenter experience. Endosc Int Open. 2015 Jun;3(3):E210-5. doi: 10.1055/s-0034-1391412. Epub 2015 Feb 27. PMID 26171433
- [Background] DeWitt J, LeBlanc J, McHenry L, Ciaccia D, Imperiale T, Chappo J, Cramer H, McGreevy K, Chriswell M, Sherman S. Endoscopic ultrasound-guided fine needle aspiration cytology of solid liver lesions: a large single-center experience. Am J Gastroenterol. 2003 Sep;98(9):1976-81. doi: 10.1111/j.1572-0241.2003.07638.x. PMID 14499774
- [Background] Hollerbach S, Willert J, Topalidis T, Reiser M, Schmiegel W. Endoscopic ultrasound-guided fine-needle aspiration biopsy of liver lesions: histological and cytological assessment. Endoscopy. 2003 Sep;35(9):743-9. doi: 10.1055/s-2003-41593. PMID 12929021
- [Background] tenBerge J, Hoffman BJ, Hawes RH, Van Enckevort C, Giovannini M, Erickson RA, Catalano MF, Fogel R, Mallery S, Faigel DO, Ferrari AP, Waxman I, Palazzo L, Ben-Menachem T, Jowell PS, McGrath KM, Kowalski TE, Nguyen CC, Wassef WY, Yamao K, Chak A, Greenwald BD, Woodward TA, Vilmann P, Sabbagh L, Wallace MB. EUS-guided fine needle aspiration of the liver: indications, yield, and safety based on an international survey of 167 cases. Gastrointest Endosc. 2002 Jun;55(7):859-62. doi: 10.1067/mge.2002.124557. PMID 12024141
- [Background] Pineda JJ, Diehl DL, Miao CL, Johal AS, Khara HS, Bhanushali A, Chen EZ. EUS-guided liver biopsy provides diagnostic samples comparable with those via the percutaneous or transjugular route. Gastrointest Endosc. 2016 Feb;83(2):360-5. doi: 10.1016/j.gie.2015.08.025. Epub 2015 Aug 22. PMID 26301407
- [Background] Sey MS, Al-Haddad M, Imperiale TF, McGreevy K, Lin J, DeWitt JM. EUS-guided liver biopsy for parenchymal disease: a comparison of diagnostic yield between two core biopsy needles. Gastrointest Endosc. 2016 Feb;83(2):347-52. doi: 10.1016/j.gie.2015.08.012. Epub 2015 Aug 13. PMID 26278654
- [Background] Gleeson FC, Clayton AC, Zhang L, Clain JE, Gores GJ, Rajan E, Smyrk TC, Topazian MD, Wang KK, Wiersema MJ, Levy MJ. Adequacy of endoscopic ultrasound core needle biopsy specimen of nonmalignant hepatic parenchymal disease. Clin Gastroenterol Hepatol. 2008 Dec;6(12):1437-40. doi: 10.1016/j.cgh.2008.07.015. Epub 2008 Jul 26. PMID 19081532
- [Background] Dewitt J, McGreevy K, Cummings O, Sherman S, Leblanc JK, McHenry L, Al-Haddad M, Chalasani N. Initial experience with EUS-guided Tru-cut biopsy of benign liver disease. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):535-42. doi: 10.1016/j.gie.2008.09.056. PMID 19231495
- [Background] Gor N, Salem SB, Jakate S, Patel R, Shah N, Patil A. Histological adequacy of EUS-guided liver biopsy when using a 19-gauge non-Tru-Cut FNA needle. Gastrointest Endosc. 2014 Jan;79(1):170-2. doi: 10.1016/j.gie.2013.06.031. Epub 2013 Jul 31. No abstract available. PMID 23916397
- [Background] Colloredo G, Guido M, Sonzogni A, Leandro G. Impact of liver biopsy size on histological evaluation of chronic viral hepatitis: the smaller the sample, the milder the disease. J Hepatol. 2003 Aug;39(2):239-44. doi: 10.1016/s0168-8278(03)00191-0. PMID 12873821
- [Background] Crawford AR, Lin XZ, Crawford JM. The normal adult human liver biopsy: a quantitative reference standard. Hepatology. 1998 Aug;28(2):323-31. doi: 10.1002/hep.510280206. PMID 9695993
- [Background] Rocken C, Meier H, Klauck S, Wolff S, Malfertheiner P, Roessner A. Large-needle biopsy versus thin-needle biopsy in diagnostic pathology of liver diseases. Liver. 2001 Dec;21(6):391-7. doi: 10.1034/j.1600-0676.2001.210605.x. PMID 11903883
- [Background] Bhatia V, Hijioka S, Hara K, Mizuno N, Imaoka H, Yamao K. Endoscopic ultrasound description of liver segmentation and anatomy. Dig Endosc. 2014 May;26(3):482-90. doi: 10.1111/den.12216. Epub 2013 Dec 19. PMID 24355092
- [Background] ASGE Standards of Practice Committee; Early DS, Acosta RD, Chandrasekhara V, Chathadi KV, Decker GA, Evans JA, Fanelli RD, Fisher DA, Fonkalsrud L, Hwang JH, Jue TL, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf RN, Shergill AK, Cash BD. Adverse events associated with EUS and EUS with FNA. Gastrointest Endosc. 2013 Jun;77(6):839-43. doi: 10.1016/j.gie.2013.02.018. No abstract available. PMID 23684089
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503

RESULTS

PARTICIPANT FLOW:
Groups:
- 19G EUS-FNA Needle First, Then 22G FNB Needle; 22G FNB Needle First, Then 19G EUS-FNA Needle: EUS-guided liver biopsy
  EUS-guided liver biopsy: Endoscopic ultrasound guided liver biopsy
  First Intervention: 10 minutes Washout: 1 minute Second Intervention: 10 minutes
Period: Overall Study
Arm/Group | 19G EUS-FNA Needle First, Then 22G FNB Needle | 22G FNB Needle First, Then 19G EUS-FNA Needle
Started | 10 (First Intervention: 10 minutes Washout: 1 minute Second Intervention: 10 minutes) | 10 (First Intervention: 10 minutes Washout: 1 minute Second Intervention: 10 minutes)
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: EUS-guided liver biopsy using a 19-gauge FNA then 22-gauge liver biopsy needle
  EUS-guided liver biopsy: Endoscopic ultrasound guided liver biopsy FNA-fine needle aspiration
Arm/Group | Total
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: mean years total population] | 50.5 (18.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex of Particpants : Male | 5
  Sex of Particpants : Female | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Specimens for Which a Histologic Diagnosis Could be Made Based Upon the Amount of Tissue Obtained With the Needle
Description: Defined by total portal structures > 5 or length of the longest piece > 15 mm) Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: 7 days
Population: specimens not particpants
Measure: Number; unit: specimens
Units Other Than Participants: specimens
Groups:
- 19 Gauge FNA: EUS-guided liver biopsy using a19-gauge liver biopsy in the left lobe
  EUS-guided liver biopsy: Endoscopic ultrasound guided liver biopsy FNA-fine needle aspiration
- 22 Gauge FNB: EUS-guided liver biopsy using a 22-gauge liver biopsy in the left lobe
  EUS-guided liver biopsy: Endoscopic ultrasound guided liver biopsy FNB-fine needle biopsy
Arm/Group | 19 Gauge FNA | 22 Gauge FNB
Number analyzed (Participants) | 20 | 20
Number analyzed (specimens) | 20 | 20
specimens | 17 | 14

2. Secondary Outcome: The Number of Specimens With a Visible Core After Needle Biopsy
Description: Presence of a visible core specimen (yes/no) Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: Day of Procedure
Population: specimens not particpants
Measure: Number; unit: specimens
Units Other Than Participants: specimens
Arm/Group | 19 Gauge FNA | 22 Gauge FNB
Number analyzed (Participants) | 20 | 20
Number analyzed (specimens) | 20 | 20
specimens | 20 | 19

3. Secondary Outcome: The Number of Specimens With a Visible Clot After Needle Biopsy
Description: Presence of visible clots in specimen (yes/no) Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: Day of Procedure
Population: specimens not participants
Measure: Number; unit: specimens
Units Other Than Participants: specimens
Arm/Group | 19 Gauge FNA | 22 Gauge FNB
Number analyzed (Participants) | 20 | 20
Number analyzed (specimens) | 20 | 20
specimens | 4 | 1

4. Secondary Outcome: The Number of Patients With Visible Bleeding After Needle Biopsy
Description: Patient with blood visible from patient's mouth, rectum with a 2 gram drop in hemoglobin Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Total Population: Adverse event evaluating the total population
Arm/Group | Total Population
Number analyzed (Participants) | 20
Participants | 0

5. Secondary Outcome: The Number of Patients With Pain 1 Day After Needle Biopsy
Description: Pain using Likert score 0-10 (10 worst) Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: 1 days
Measure: Count of Participants; unit: Participants
Groups:
- Total Population: Adverse events evaluating the total population
Arm/Group | Total Population
Number analyzed (Participants) | 20
Participants | 0

6. Secondary Outcome: The Number of Patients With Pain 7 Day After Needle Biopsy
Description: as for outcome 5
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Total Population
Number analyzed (Participants) | 20
Participants | 1

7. Secondary Outcome: The Number of Patients Requiring Medical Care After Needle Biopsy
Description: Patient requiring visit to healthcare center (emergency room, hospital, call to service) within time 7 days Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: 7 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Total Population
Number analyzed (Participants) | 20
Participants | 1

8. Secondary Outcome: Number of Portal Tracts (PT) in the Specimen (Total) Under Histologic Examination
Description: Number of portal tracts (PT) in the specimen (total) under histologic examination Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: 7 days
Population: specimens not participants
Measure: Mean (Standard Deviation); unit: mean portal tracts
Units Other Than Participants: specimens
Groups:
- 19 Gauge FNA: EUS-guided liver biopsy using a19-gauge liver biopsy in the left lobe
  EUS-guided liver biopsy: Endoscopic ultrasound guided liver biopsy
- 22 Gauge FNB: EUS-guided liver biopsy using a 22-gauge liver biopsy in the left lobe
  EUS-guided liver biopsy: Endoscopic ultrasound guided liver biopsy
Arm/Group | 19 Gauge FNA | 22 Gauge FNB
Number analyzed (Participants) | 20 | 20
Number analyzed (specimens) | 20 | 20
mean portal tracts | 7.4 (5.9) | 6.1 (7.2)

9. Secondary Outcome: Aggregate Specimen Length Under Histologic Examination
Description: Length of all the tissue (centimeters) by adding the sum of all pieces Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: 7 days
Population: specimens not participants
Measure: Mean (Standard Deviation); unit: cm for portal tracts of specimens
Units Other Than Participants: specimens
Arm/Group | 19 Gauge FNA | 22 Gauge FNB
Number analyzed (Participants) | 20 | 20
Number analyzed (specimens) | 20 | 20
cm for portal tracts of specimens | 76.5 (35.4) | 66.9 (47.8)

10. Secondary Outcome: Length of the Longest Piece Under Histologic Examination
Description: length of the longest tissue biopsy piece (centimeters) as measured by pathology Subjects underwent a left liver biopsy using a 19-gauge FNA needle, 22-gauge FNB needle, right liver biopsies also using the 19-gauge FNA and 22-gauge FNB.
  FNA-fine needle aspiration FNB-fine needle biopsy
Time Frame: 7 days
Population: specimens not participants
Measure: Mean (Standard Deviation); unit: mean cm for portal tracts of specimens
Units Other Than Participants: specimens
Arm/Group | 19 Gauge FNA | 22 Gauge FNB
Number analyzed (Participants) | 20 | 20
Number analyzed (specimens) | 20 | 20
mean cm for portal tracts of specimens | 13.2 (5.1) | 10.8 (6.8)

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Total Population: EUS-guided liver biopsy using 19 g needle and 22 g needle in a cross-over design. Results were evaluated for groups undergoing 19 g needle followed by 22 g needle and 22 g needle followed by 19 g needle.
  EUS-guided liver biopsy: Endoscopic ultrasound guided liver biopsy
  NOTE that as this is a cross-over design adverse events were reported occurred were reported on a per-patient basis. Given that events were reported after the procedure, unique to each patient, and cannot be expressed based upon a per-intervention basis as both interventions were performed on each patient and only one patient can have one unique intervention which is impossible to determine the route-source intervention as the culprit due to cross-over design same session.
Arm/Group | Total Population
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
No blinding, single-center, no generalization to community, carrier effect with cross-over design, obesity, second pass.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT02967991/Prot_000.pdf
  • Informed Consent Form (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT02967991/ICF_001.pdf
  • Statistical Analysis Plan (2016-08-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02967991/SAP_002.pdf